CLINICAL TRIAL: NCT02768727
Title: A Test of Neural Inertia in Humans With Xenon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 824229
Record Dates: First submitted 2016-04-15; First posted 2016-05-11 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Neurocognitive Dysfunction
Keywords: neurocognitive function; neural inertia; xenon gas
MeSH Terms: conditions — Cognition Disorders | interventions — Xenon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xenon (Experimental): Xenon anesthesia to determine if neural inertia is present in humans as visualized by CT imaging.
  Interventions: Drug: Xenon

INTERVENTIONS:
Drug: Xenon — drug given in concentrations of 0% to 60% over period of 2 hours

SUMMARY:
The dual objectives of this study are to determine if the phenomenon of neural inertia is present in humans and to determine whether the order of neurocognitive function is invariant among anesthetic agents. This study will enroll 24 healthy volunteers, ages 20-40 years, who will receive xenon gas (concentrations ranging from 0% to 60%) delivered via inhaled route through the ENHANCER 3000.

DETAILED DESCRIPTION:
This is a multimodal, nonrandomized study of healthy subjects. After meeting enrollment criteria, subjects will receive a baseline neurocognitive testing on a computer for 15 minutes and will then receive a wrist watch actigraphy device to record their rest/activity patterns over 8-14 days. On the study day (roughly two weeks later), repeat baseline neurocognitive testing will be performed after subjects are fitted with a high density EEG head cap. The actual intervention (delivery of inhaled xenon gas in stepwise increasing followed by decreasing doses) should occur over 2 hours along with verbal tests to assess the presence/absence of consciousness at each xenon concentration. Xenon doses have been chosen specifically to evaluate the point at which individuals lose and then regain consciousness. Doses are escalated up through those used in human anesthesiology (75%) that permit surgery. After exposure, serial neurocognitive testing will occur every 30 minutes for 3 hours post emergence. Subjects are discharged from the study's intervention day to home only upon reaching standard post-anesthesia care unit criteria (modified Aldrete score ≥9). A post-procedure follow up phone call will occur within 24 hours of anesthetic exposure to ensure that the subject remains well. The individual's involvement is completed upon returning the Actigraphy watch 1 week after the exposure day. The expected duration of subject participation is 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ages 20-40 years old
* American Society of Anesthesiologists (ASA) Physical Status I or II (i.e. healthy)
* Body Mass Index <30 kg/m2
* Easily visible uvula

Exclusion Criteria:

* Any physical signs that would suggest a difficult airway (e.g. mouth opening <3cm, short distance between the chin and neck, poor mandibular subluxation, thick neck)
* History of reactive airway disease
* Current or history of neuropsychiatric disorders
* History or current use of psychotropic medications,
* History or current obstructive sleep apnea
* Current or history of cardiovascular disease or arrhythmias,
* Current or history of chronic sleep disorders
* History of postoperative nausea/vomiting
* Family history of problems with anesthesia (including but not limited to malignant hyperthermia),
* Current or history of Motion sickness
* Current tobacco use
* Current pregnancy or currently breastfeeding
* Positive urine toxicology screen
* History of seizure disorder, head injury, or brain tumor
* Alcohol consumption greater than 12 drinks per week or more than 4 drinks on any single day
* Inability to provide informed consent
* Inability to achieve mask seal on intervention day

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04; Primary Completion 2019-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
xenon concentrations at which consciousness is lost and regained | 4 hours
  To determine in healthy human volunteers if the brain concentrations of xenon (as determined by CT imaging) are identical at the point of loss and return of consciousness.

SECONDARY OUTCOMES:
Neurocognitive recovery upon emergence from xenon as measured by neurocognitive battery testing | 4 hours
  To determine if the order of neurocognitive recovery upon emergence from xenon general anesthesia is sequential or simultaneous and if the former is true to determine if the pattern is identical to that of isoflurane (as measured in a previously completed study).
Effects of xenon on gross motor activity as measured by actigraphy | 3 weeks
  To determine if xenon induces transient phase shifts in rest-activity rhythms (as measured from actigraphy) as has been previously reported for isoflurane.
Effects of xenon on brain electrical activity as measured by EEG | 4 hours
  To determine effects of xenon on brain electrical activity corresponding to loss and subsequent return of consciousness and also at points corresponding to return as each neurocognitive domain returns to its baseline following exposure to xenon as measured by electroencephalogram (EEG).

CONTACTS AND LOCATIONS:
Overall Officials: Maz B Kelz, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No